CLINICAL TRIAL: NCT03187093
Title: Cognitive Dysfunction in Patients With Major Depressive Disorder, Clinical Peculiarities, Biological Markers, and Treatment Efficacy
Brief Title: Cognitive Dysfunction in MDD Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oleg Levada (Other)
Responsible Party: Sponsor-Investigator, Oleg Levada, MD, ScD (psychiatry), PhD (neurology), Psychiatry course chief, State Institution, Zaporizhzhia Medical Academy of Post-Graduate Education Ministry of Health of Ukraine
Organization: State Institution, Zaporizhzhia Medical Academy of Post-Graduate Education Ministry of Health of Ukraine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11031215
Record Dates: First submitted 2017-06-01; First posted 2017-06-14 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Vortioxetine; Cognitive dysfunction; IGF-1; BDNF; Functioning
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction | interventions — Vortioxetine; Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vortioxetine (Active Comparator)
  Interventions: Drug: Vortioxetine
- Escitalopram (Active Comparator)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Vortioxetine — 10-20 mg once daily for 8 weeks
  Other Names: Brintellix; Trintellix
  Arms: Vortioxetine
Drug: Escitalopram — 10-20 mg once daily for 8 weeks
  Arms: Escitalopram

SUMMARY:
Major Depressive Disorder (MDD) is one of the most prevalent mental diagnosis within the worldwide population. Although there is evidence about relationship between MDD and cognitive dysfunction, still the correlations between biomarkers and the severity of the disorder or the level of cognitive dysfunction need further research. Therefore, the aim of the study is to determine such relationships in Ukrainian population.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient 18 to 65 years of age
* Meets DSM-5 criteria for MDD
* Depressive episode duration ≥ 2 months
* The participant has MARDS total score ≥ 7
* Free of psychotropic medications for at least 5 half-lives before baseline
* Fluent in Russian/Ukrainian

Exclusion Criteria:

* Current diagnosis or history of manic/hypomanic episode
* Any other psychiatric diagnosis that is considered the primary diagnosis
* Any significant personality disorder diagnosis
* High suicidal risk, defined by clinician judgment
* Substance dependence/abuse in the past year
* Significant neurological disorders, head trauma, or other unstable medical conditions
* History of endocrinological diseases
* Pregnant or breastfeeding
* Psychosis in the current episode
* High risk for hypomanic switch
* Cognitive or language impairment of such severity as to adversely affect the performance of tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to week 8 in Sheehan Disability Scale | Baseline to Week 8

SECONDARY OUTCOMES:
Change from baseline to week 8 in MADRS | Baseline to Week 8
Change from baseline to week 8 in PHQ-9 | Baseline to Week 8
Change from baseline to week 8 in CGI-S | Baseline to Week 8
Change from baseline to week 8 in PDQ-5-D | Baseline to Week 8
Change from baseline to week 8 in RAVLT | Baseline to Week 8
Change from baseline to week 8 in TMT-B | Baseline to Week 8
Change from baseline to week 8 in DSST | Baseline to Week 8
Change from baseline to week 8 in plasma levels of IGF-1 | Baseline to Week 8
Change from baseline to week 8 in plasma levels of BDNF | Baseline to Week 8
Change from baseline to week 8 in plasma levels of CRP | Baseline to Week 8
Change from baseline to week 8 in plasma levels of cortisol | Baseline to Week 8
Change from baseline to week 8 in plasma levels of ACTH | Baseline to Week 8

CONTACTS AND LOCATIONS:
Locations (1):
- State Institution "Zaporizhzhia Medical Academy of Postgraduate Education Ministry of Health of Ukraine", Zaporizhzhia, Ukraine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Levada OA, Troyan AS, Pinchuk IY. Serum insulin-like growth factor-1 as a potential marker for MDD diagnosis, its clinical characteristics, and treatment efficacy validation: data from an open-label vortioxetine study. BMC Psychiatry. 2020 May 8;20(1):208. doi: 10.1186/s12888-020-02636-7. PMID 32384884